CLINICAL TRIAL: NCT02152319
Title: PDRemote Phase II: Automated Telehealth Diagnostics for Remote Parkinson Monitoring
Brief Title: Automated Telehealth Diagnostics for Remote Parkinson Monitoring
Acronym: PDRemote
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: University of Rochester (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R44MD004049 (NIH); 5R44MD004049-05 (NIH)
Record Dates: First submitted 2014-05-27; First posted 2014-06-02 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Telemedicine; Telehealth; Kinesia; Tremor; Bradykinesia; Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Tremor; Hypokinesia; Dyskinesias | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- KHV reporting (Experimental): Clinicians will view the motor symptom severity reports and videoconference to titrate medications.
  Interventions: Device: KHV reporting; Procedure: Standard care
- Standard care (Active Comparator): Subjects in this group will still use KHV at home to minimize any placebo effects that could be attributed to using the system; however, clinicians will view the motor symptom severity reports and videoconference to titrate medications solely for the experimental subjects.
  Interventions: Procedure: Standard care

INTERVENTIONS:
Device: KHV reporting — Clinicians will view the KHV motor symptom severity reports and use KHV to videoconference with subjects to titrate medications.
  Other Names: Kinesia HomeView
  Arms: KHV reporting
Procedure: Standard care — Subjects will receive the same disease management as if they were not participating in this study.

SUMMARY:
The objective is to clinically assess the Kinesia HomeView system for automated and remote monitoring of Parkinson's disease (PD) motor symptoms.

DETAILED DESCRIPTION:
Currently, there is limited access to movement disorder specialist centers for a significant portion of the PD population. Treatment effectiveness is judged during office visits by improvement of patient motor symptoms and quality of life. Clinicians evaluate patients by having them perform specific motor tasks and rating the severity on a 0-4 scale. A major limitation is that a single evaluation in a clinical setting may not accurately reflect motor symptom fluctuations experienced over the course of a day, week, or month. Clinicians currently lack effective, affordable medical devices that can be easily delivered to a patient's home for monitoring symptoms on a more continuous basis as motor symptoms typically change throughout the day. Kinesia HomeView provides a repeatable, automated system clinicians can use to remotely monitor PD motor symptoms on a more continuous basis in a patient's home. The investigators hypothesize use of the Kinesia HomeView system will improve outcomes and decrease costs especially for patient populations in areas not in close proximity to movement disorder specialists.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with self-reported clinically-confirmed diagnosis of idiopathic Parkinson disease.
* Be fluent in English
* Willing and able to provide informed consent

Exclusion Criteria:

* Inability to carry out study activities
* Subjects with cognitive deficits that would prevent following instructions and serious medical conditions that would compromise a subject's safety
* Subjects who have dementia, exhibited by those with a score less than 22 on the Montreal Cognitive Assessment (MoCA)
* Subjects with deep brain stimulation (DBS)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percent of subjects completing remote assessments | 7 Months
  Percent of subjects who successfully completed the requested home-based Kinesia HomeView (KHV) automated motor assessments.

SECONDARY OUTCOMES:
Percent of remote assessments completed | 7 Months
  Percent of remote home-based Kinesia-HomeView automated motor assessments successfully completed .
KHV Motor Scores | 7 Months
  Tremor, bradykinesia, and dyskinesia scores given by the KHV system.
KHV measured fluctuations | 7 Months
  Changes in KHV motor scores throughout each day.
PDQ-39 responses | 7 Months
  PDQ-39 quality of life survey responses.
PACIC responses | 7 Months
  The Patient Assessment of Care for Chronic Conditions (PACIC) is a questionnaire that measures specific actions or qualities of care
PAM-13 responses | 7 Months
  The Patient Activation Measure (PAM) assessment gauges the knowledge, skills and confidence essential to managing one's own health and healthcare.
Number of clinic visits | 7 Months
Number of patient/clinician communications | 7 Months
Number and type of medication changes | 7 Months
Number of videoconferences completed | 7 Months
Unified Parkinson's Disease Rating Scale (UPDRS) | 7 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Giuffrida, Ph.D., Principal Investigator — Great Lakes NeuroTechnologies; Dustin A Heldman, Ph.D., Study Director — Great Lakes NeuroTechnologies
Locations (1):
- University of Rochester, Rochester, New York, United States